CLINICAL TRIAL: NCT01518777
Title: Reducing Radioisotope Dose in Regadenoson SPECT Myocardial Perfusion Imaging: Comparison of Half-Dose Scans Using a Novel Solid-State-Detector Dedicated Cardiac Camera to Full Dose Scans Acquired On Standard Equipment
Brief Title: Reducing Radioisotope Dose: the Half-Dose CZT Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S.M.Chang, MD (Other)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor-Investigator, S.M.Chang, MD, Sponsor-Investigator/Principal Investigator, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00006818
Record Dates: First submitted 2012-01-23; First posted 2012-01-26 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Half-dose isotope for NuclearStressTest (Other): Intervention is Nuclear stress test of the heart. Single-arm of this study "Half-dose of isotope for Nuclear stress test" is group of study subjects who will do Research Nuclear stress test with half-dose of isotope that normally used for routine Nuclear stress test. Isotope is the tracer CZT (cadmium zinc telluride) that used for Nuclear stress test routinely to see the function of arteries of the heart. Patients with suspected Coronary Artery Disease who meet entry criteria undergo a research nuclear stress test using a decreased dose of isotope, using a new camera.
  Interventions: Other: Half-dose isotope for NuclearStressTest

INTERVENTIONS:
Other: Half-dose isotope for NuclearStressTest — Half-dose of tracer or radioisotope will be used for Nuclear stress test of the heart. This is imaging test of the heart to see the function of arteries of the heart.
  Other Names: SPECT using CZT

SUMMARY:
This is a pilot study to see whether cardiac imaging can be performed using half the standard dose of radioisotope.

DETAILED DESCRIPTION:
The aim of this study is to compare the image quality of the half radioisotope dose scans obtained using a CZT (cadmium zinc telluride) camera with scans acquired using a standard of care imaging protocol/radioisotope dose performed on a traditional (conventional) camera.

The proposed strategy of a half dose/extended time protocol with the CZT camera should yield a similar count activity and consequently image quality equivalent to that detected by a conventional SPECT system.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age and referred for a clinically-indicated stress SPECT MPI study
* suspected or known coronary artery disease
* written informed consent

Exclusion Criteria:

* Evidence of a normal baseline scan after at least 50% of the protocol acquired baseline scans have been interpreted as being normal
* Participation in another investigational study within the preceding month
* Pregnant and/or breast-feeding female
* ECG evidence of left bundle branch block or paced rhythm
* Evidence of non-ischemic cardiomyopathy
* Presence of hypertrophic cardiomyopathy and/or severe valvular heart disease
* Severe claustrophobia or inability to lie flat for 20 minutes (the anticipated amount of time to complete the procedure)
* Known allergy to technetium-99m
* Potential contraindications to regadenoson use, due to severe lung disease; severe bradycardia (heart rate < 40 beats/min); second- or third degree atrioventricular heart block; sick sinus syndrome; long QT syndrome; severe hypotension; or decompensated heart failure.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-01; Primary Completion 2016-12-16 (Actual); Study Completion 2016-12-16 (Actual)

PRIMARY OUTCOMES:
Image quality of the half-dose CZT versus full dose scans | 1 Week

SECONDARY OUTCOMES:
Total radiation dose/exposure of the half-dose CZT vs. full dose scans | 1 Week
Total myocardial count activity and count rates obtained during each scan | 1 Week
Agreement between the half-dose CZT vs. full dose scans on the presence and extent of fixed or reversible defects on a per-patient and vessel basis | 1 Week
Agreement between the half-dose vs. full dose scans on gated data such as EF, left ventricular (LV) end-diastolic volume, LV end-systolic volume | 1 Week

CONTACTS AND LOCATIONS:
Overall Officials: Su Min Chang, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
No.

REFERENCES:
- [Background] Shaw LJ, Iskandrian AE. Prognostic value of gated myocardial perfusion SPECT. J Nucl Cardiol. 2004 Mar-Apr;11(2):171-85. doi: 10.1016/j.nuclcard.2003.12.004. No abstract available. PMID 15052249
- [Background] Henzlova MJ, Cerqueira MD, Mahmarian JJ, Yao SS; Quality Assurance Committee of the American Society of Nuclear Cardiology. Stress protocols and tracers. J Nucl Cardiol. 2006 Nov;13(6):e80-90. doi: 10.1016/j.nuclcard.2006.08.011. No abstract available. PMID 17174798
- [Background] Einstein AJ, Moser KW, Thompson RC, Cerqueira MD, Henzlova MJ. Radiation dose to patients from cardiac diagnostic imaging. Circulation. 2007 Sep 11;116(11):1290-305. doi: 10.1161/CIRCULATIONAHA.107.688101. No abstract available. PMID 17846343
- [Background] Einstein AJ, Henzlova MJ, Rajagopalan S. Estimating risk of cancer associated with radiation exposure from 64-slice computed tomography coronary angiography. JAMA. 2007 Jul 18;298(3):317-23. doi: 10.1001/jama.298.3.317. PMID 17635892
- [Background] Fazel R, Krumholz HM, Wang Y, Ross JS, Chen J, Ting HH, Shah ND, Nasir K, Einstein AJ, Nallamothu BK. Exposure to low-dose ionizing radiation from medical imaging procedures. N Engl J Med. 2009 Aug 27;361(9):849-57. doi: 10.1056/NEJMoa0901249. PMID 19710483
- [Background] Fazel R, Shaw LJ. Radiation exposure from radionuclide myocardial perfusion imaging: concerns and solutions. J Nucl Cardiol. 2011 Aug;18(4):562-5. doi: 10.1007/s12350-011-9403-y. No abstract available. PMID 21638151
- [Background] Herzog BA, Buechel RR, Katz R, Brueckner M, Husmann L, Burger IA, Pazhenkottil AP, Valenta I, Gaemperli O, Treyer V, Kaufmann PA. Nuclear myocardial perfusion imaging with a cadmium-zinc-telluride detector technique: optimized protocol for scan time reduction. J Nucl Med. 2010 Jan;51(1):46-51. doi: 10.2967/jnumed.109.065532. Epub 2009 Dec 15. PMID 20008999
- [Background] Buechel RR, Herzog BA, Husmann L, Burger IA, Pazhenkottil AP, Treyer V, Valenta I, von Schulthess P, Nkoulou R, Wyss CA, Kaufmann PA. Ultrafast nuclear myocardial perfusion imaging on a new gamma camera with semiconductor detector technique: first clinical validation. Eur J Nucl Med Mol Imaging. 2010 Apr;37(4):773-8. doi: 10.1007/s00259-009-1375-7. Epub 2010 Jan 27. PMID 20107783
- [Background] Esteves FP, Raggi P, Folks RD, Keidar Z, Askew JW, Rispler S, O'Connor MK, Verdes L, Garcia EV. Novel solid-state-detector dedicated cardiac camera for fast myocardial perfusion imaging: multicenter comparison with standard dual detector cameras. J Nucl Cardiol. 2009 Nov-Dec;16(6):927-34. doi: 10.1007/s12350-009-9137-2. Epub 2009 Aug 18. PMID 19688410
- [Background] Gimelli A, Bottai M, Giorgetti A, Genovesi D, Kusch A, Ripoli A, Marzullo P. Comparison between ultrafast and standard single-photon emission CT in patients with coronary artery disease: a pilot study. Circ Cardiovasc Imaging. 2011 Jan;4(1):51-8. doi: 10.1161/CIRCIMAGING.110.957399. Epub 2010 Nov 10. PMID 21068188
- [Background] Duvall WL, Croft LB, Ginsberg ES, Einstein AJ, Guma KA, George T, Henzlova MJ. Reduced isotope dose and imaging time with a high-efficiency CZT SPECT camera. J Nucl Cardiol. 2011 Oct;18(5):847-57. doi: 10.1007/s12350-011-9379-7. Epub 2011 Apr 29. PMID 21528422
- [Background] Duvall WL, Sweeny JM, Croft LB, Barghash MH, Kulkarni NK, Guma KA, Henzlova MJ. Comparison of high efficiency CZT SPECT MPI to coronary angiography. J Nucl Cardiol. 2011 Aug;18(4):595-604. doi: 10.1007/s12350-011-9382-z. Epub 2011 Jun 3. PMID 21638154
- [Background] Mahmarian JJ, Shaw LJ, Olszewski GH, Pounds BK, Frias ME, Pratt CM; INSPIRE Investigators. Adenosine sestamibi SPECT post-infarction evaluation (INSPIRE) trial: A randomized, prospective multicenter trial evaluating the role of adenosine Tc-99m sestamibi SPECT for assessing risk and therapeutic outcomes in survivors of acute myocardial infarction. J Nucl Cardiol. 2004 Jul-Aug;11(4):458-69. doi: 10.1016/j.nuclcard.2004.05.003. PMID 15295415
- [Background] ICRP. Radiation dose to patients from radiopharmaceuticals. Addendum 3 to ICRP Publication 53. ICRP Publication 106. Approved by the Commission in October 2007. Ann ICRP. 2008;38(1-2):1-197. doi: 10.1016/j.icrp.2008.08.003. PMID 19154964
- [Background] The 2007 Recommendations of the International Commission on Radiological Protection. ICRP publication 103. Ann ICRP. 2007;37(2-4):1-332. doi: 10.1016/j.icrp.2007.10.003. PMID 18082557
- [Background] Radiation dose to patients from radiopharmaceuticals (addendum 2 to ICRP publication 53). Ann ICRP. 1998;28(3):1-126. doi: 10.1016/s0146-6453(99)00006-8. PMID 10840563